CLINICAL TRIAL: NCT02724709
Title: Semi-automatic assessMent of Aortic Roots by Three-dimensional transoEsophageal echocaRdiography (SMARTER)
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Principal Investigator, Bin Lu, Professor and Director of Radiologic Imaging, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2016-096
Record Dates: First submitted 2016-03-21; First posted 2016-03-31 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Aortic Valve Disease
Keywords: Automatic Data Processing; Three-Dimensional Echocardiography; Aortic Valve
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Three-dimensional transoesophageal echocardiography — Three-dimensional transoesophageal echocardiography, analysed by eSie valve software (Siemens)
Procedure: Computed tomography — Computed tomography, analysed by Synovia Workstation (Siemens)

SUMMARY:
The progress in surgery of the aortic root and the evolution of transcatheter aortic valve replacement as an alternative to surgical treatment in selected patients have refocused the need for quantitative imaging of the aortic root during transcatheter aortic valve replacement and valve-sparing aortic root surgery. In this study, we aim to assess the ability of semi-automated quantitative modeling (eSie Valves, Autovalve prototype version, Siemens Medical Solutions, USA) of the aortic valve and root in patients with clinical normal aortic valve and root, who are indicated for both 3D transesophageal echocardiography (TEE) and computed tomographic (CT) due to atrial fibrillation or patent foramen ovale. Measures of the aortic valve and root obtained by 2D TEE, 3D TEE and CT are compared, and the ability of the semi-automated 3D TEE modeling software is tested. Given the workflow advantages of automation, this 3D TEE approach may enhance the clinical adoption of routine 3-dimensional imaging beyond CT.

DETAILED DESCRIPTION:
Recent developments in aortic root interventions have focused on the need for 3-dimensional imaging of the aortic functional anatomy. The progress in surgery of the aortic root and the evolution of transcatheter aortic valve replacement as an alternative to surgical treatment in selected patients have refocused the need for quantitative imaging of the aortic root during transcatheter aortic valve replacement and valve-sparing aortic root surgery. In this study, we aim to assess the ability of semi-automated quantitative modeling (eSie Valves, Autovalve prototype version, Siemens Medical Solutions, USA) of the aortic valve and root in patients with clinical normal aortic valve and root, who are indicated for both 3D transesophageal echocardiography (TEE) and computed tomographic (CT) due to atrial fibrillation or patent foramen ovale. Measures of the aortic valve and root obtained by 2D TEE, 3D TEE and CT are compared, and the ability of the semi-automated 3D TEE modeling software is tested. Given the workflow advantages of automation, this 3D TEE approach may enhance the clinical adoption of routine 3-dimensional imaging beyond CT.

ELIGIBILITY:
Inclusion Criteria:

* both transesophageal echocardiography (TEE) and computed tomographic (CT) are referred by cardiologists
* apparent normal aortic valve and root structure
* written consent

Exclusion Criteria:

* post-operation of aortic valve
* severe cardiomyopathy
* cardiac functional insufficiency (NYHA III or IV)
* contraindications for either TEE or cardiac CT angiography

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical normal aortic valve and root, who are indicated for both transesophageal echocardiography (TEE) and computed tomographic (CT) due to atrial fibrillation or patent foramen ovale.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Accuracy | Through study completion, an average of 1 month
  Compare semi-automatic assessment of 3D TEE to CT measurement

SECONDARY OUTCOMES:
Cost | Through study completion, an average of 1 month
  Compare cost between 3D TEE and CT
Labor time | Through study completion, an average of 1 month
  Compare labor time between 3D TEE and CT

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wang, M.D., Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Garcia-Martin A, Lazaro-Rivera C, Fernandez-Golfin C, Salido-Tahoces L, Moya-Mur JL, Jimenez-Nacher JJ, Casas-Rojo E, Aquila I, Gonzalez-Gomez A, Hernandez-Antolin R, Zamorano JL. Accuracy and reproducibility of novel echocardiographic three-dimensional automated software for the assessment of the aortic root in candidates for thanscatheter aortic valve replacement. Eur Heart J Cardiovasc Imaging. 2016 Jul;17(7):772-8. doi: 10.1093/ehjci/jev204. Epub 2015 Aug 27. PMID 26320167
- [Background] Calleja A, Thavendiranathan P, Ionasec RI, Houle H, Liu S, Voigt I, Sai Sudhakar C, Crestanello J, Ryan T, Vannan MA. Automated quantitative 3-dimensional modeling of the aortic valve and root by 3-dimensional transesophageal echocardiography in normals, aortic regurgitation, and aortic stenosis: comparison to computed tomography in normals and clinical implications. Circ Cardiovasc Imaging. 2013 Jan 1;6(1):99-108. doi: 10.1161/CIRCIMAGING.112.976993. Epub 2012 Dec 10. PMID 23233743
- [Background] Chambers JB, Myerson SG, Rajani R, Morgan-Hughes GJ, Dweck MR. Multimodality imaging in heart valve disease. Open Heart. 2016 Mar 8;3(1):e000330. doi: 10.1136/openhrt-2015-000330. eCollection 2016. PMID 26977308
- [Background] Hahn RT, Little SH, Monaghan MJ, Kodali SK, Williams M, Leon MB, Gillam LD. Recommendations for comprehensive intraprocedural echocardiographic imaging during TAVR. JACC Cardiovasc Imaging. 2015 Mar;8(3):261-287. doi: 10.1016/j.jcmg.2014.12.014. PMID 25772834
- [Derived] Zhang M, Wan L, Liu K, Wu W, Li H, Wang Y, Lu B, Wang H. Aortic roots assessment by an automated three-dimensional transesophageal echocardiography: an intra-individual comparison. Int J Cardiovasc Imaging. 2019 Nov;35(11):2029-2036. doi: 10.1007/s10554-019-01664-z. Epub 2019 Jul 11. PMID 31297671